CLINICAL TRIAL: NCT02412566
Title: Compassionate Use of an Intravenous Fat Emulsion Comprised of Soy Oil, Medium Chain Triglycerides, Olive Oil, and Fish Oil for Children With Parenteral Nutrition Induced Liver Injury
Brief Title: SMOF Lipid for Children With Parenteral Nutrition Induced Liver Injury
Acronym: SMOF
Status: Approved for marketing | Type: Expanded Access
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Muralidhar Premkumar, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-34444
Record Dates: First submitted 2015-03-25; First posted 2015-04-09 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cholestasis; Growth Failure
Keywords: cholestasis; growth failure; intravenous fat emulsion; SMOF
MeSH Terms: conditions — Cholestasis; Failure to Thrive | interventions — SMOFlipid

INTERVENTIONS:
Drug: SMOFlipid — Therapy with SMOFlipid will be provided at a targeted dose of 3 gm/kg/day (by continuous infusion). SMOFlipid will be initiated and advanced according to the following guidelines: Day 1 - provide 1 g/kg; Day 2 - provide 2 g/kg; Day 3 - provide 3 g/kg. SMOFlipid will be infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition.
  Other Names: SMOF

SUMMARY:
While fish-oil lipid emulsions have shown a benefit to the treatment of parenteral nutrition (PN)-associated cholestasis, the dose is limited to 1 g/kg/day. Similarly, in early PN-associated cholestasis the dose of soy-based lipid is limited to 1 g/kg/day. Often the calories that are lost from this relative decreased dose of lipids can be provided by adjusting the dextrose content of the PN solution and providing a higher glucose infusion rate. In some cases, this is not tolerated or even with maximizing this strategy, growth is inadequate. Inadequate growth is a direct cause of poor outcomes including poorer neurological outcome, failure to be able to stop mechanical ventilation and poorer growth of their often already damaged intestine. These outcomes can lead to severe disability and death. Therefore, infants receiving only 1 g/kg/day of lipids who are not adequately growing must have a greater intake of lipids to meet their needs for weight, length, and head circumference growth.

SMOFlipid (Fresenius Kabi, Bad Homburg, Germany) contains a mixture of 4 different lipid sources: soybean oil providing essential fatty acids, olive oil rich in monounsaturated fatty acids which are less susceptible to lipid peroxidation than polyunsaturated fatty acids, medium-chain triglycerides showing a faster metabolic clearance than long-chain triglycerides, and fish oil for the supply of omega-3 fatty acids. It is safe to give in what is the usual dose for lipid therapy in neonates of 3 g/kg/day, rather than being limited to 1 g/kg/day as we do with cholestatic infants receiving Omegaven or soy lipids. Because this product includes both omega-6 and omega-3 lipids, it provides the benefits of the omega-3s for the liver and provides more than enough omega-6s to meet essential fatty acid requirements. Its use in situations in which growth is inadequate in babies who must be restricted to 1 g/kg/day can be expected to improve their growth and likely markedly increase their chances of both a good neurological outcome and survival.

Purpose: We want to find out if this new intravenous fat mixture (SMOFlipid) will help promote good growth while reducing the severity (or seriousness) of liver disease or help put an end to liver disease in infants.

DETAILED DESCRIPTION:
Therapy with SMOFlipid will be provided at a targeted dose of 3 gm/kg/day (by continuous infusion). SMOFlipid will be initiated and advanced according to the following guidelines: Day 1 - provide 1 g/kg; Day 2 - provide 2 g/kg; Day 3 - provide 3 g/kg. SMOFlipid will be infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition. The same standards of care provided to all patients receiving parenteral nutrition (PN) solution will be followed.

Essential fatty acid levels will be measured at 4 and 12 weeks after the initiation of SMOFlipid. This time frame will be used to assess essential fatty acids of both inpatients and outpatients. These labs are clinically indicated; therefore, we will record the results of the total fatty acid lipid profile panel from the medical record into our case report forms.

Patients will remain on SMOFlipid until weaned from PN. In the event that a patient who has been listed for a liver or liver/intestinal transplant has an organ become available, the participation in this protocol will not preclude them from receiving the transplant. SMOFlipid will not be administered post transplant.

If the infant no longer is requiring any PN, then the SMOFlipid will be stopped regardless of bilirubin. If the bilirubin is less than 2 mg/dL but the child still requires PN, then the SMOFlipid will be continued up until the infant no longer requires PN. The reason for stopping SMOFlipid when the infant no longer requires PN is that this would be the only reason many infants would still need IV access and therefore the risk of maintaining IV access only for the medication is likely to exceed the benefit of SMOFlipid at that point.

Babies who receive SMOFlipid are not precluded from receiving Omegaven per that compassionate use protocol (H-23365) if they meet the inclusion criteria for that protocol.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 14 days old and less than 1 year of age.
* Greater than 1.5 kg.
* Mild cholestasis, defined as a conjugated bilirubin between 0.5-1.9 mg/dL, or currently receiving Omegaven (fish oil lipid emulsion) with a conjugated bilirubin between 0.0-1.9 mg/dL.
* Currently receiving 1 g/kg/day of either Omegaven (H-23365) or soy-based Intralipid (standard therapy)
* Evidence of growth of weight, head circumference or length below our standards for post-menstrual age for at least 1 week.
* Be expected to require intravenous nutrition for at least an additional 21 days.

Exclusion Criteria:

* Have a congenitally lethal condition (e.g. Trisomy 13).
* Have clinically severe bleeding or clinical liver failure not able to be managed with routine measures.
* Have evidence of a viral hepatitis or primary liver disease as the primary etiology of their cholestasis.
* Have other health problems such that survival is extremely unlikely even if the infant's cholestasis improves

Ages: 14 Days to 1 Year | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Muralidhar H. Premkumar, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine / Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Rayyan M, Devlieger H, Jochum F, Allegaert K. Short-term use of parenteral nutrition with a lipid emulsion containing a mixture of soybean oil, olive oil, medium-chain triglycerides, and fish oil: a randomized double-blind study in preterm infants. JPEN J Parenter Enteral Nutr. 2012 Jan;36(1 Suppl):81S-94S. doi: 10.1177/0148607111424411. PMID 22237883
- [Background] Goulet O, Antebi H, Wolf C, Talbotec C, Alcindor LG, Corriol O, Lamor M, Colomb-Jung V. A new intravenous fat emulsion containing soybean oil, medium-chain triglycerides, olive oil, and fish oil: a single-center, double-blind randomized study on efficacy and safety in pediatric patients receiving home parenteral nutrition. JPEN J Parenter Enteral Nutr. 2010 Sep-Oct;34(5):485-95. doi: 10.1177/0148607110363614. PMID 20852176
- [Background] Tomsits E, Pataki M, Tolgyesi A, Fekete G, Rischak K, Szollar L. Safety and efficacy of a lipid emulsion containing a mixture of soybean oil, medium-chain triglycerides, olive oil, and fish oil: a randomised, double-blind clinical trial in premature infants requiring parenteral nutrition. J Pediatr Gastroenterol Nutr. 2010 Oct;51(4):514-21. doi: 10.1097/MPG.0b013e3181de210c. PMID 20531018
- See also: Children's Nutrition Research Center — https://www.bcm.edu/departments/pediatrics/sections-divisions-centers/childrens-nutrition-research-center/